CLINICAL TRIAL: NCT00230477
Title: Efficacy of Adefovir Dipivoxil Versus Adefovir Dipivoxil Plus Lamivudine for the Treatment of Chronic Hepatitis B in Patients With Normal Baseline ALT
Brief Title: Hepsera Versus Hepsera Plus Lamivudine for Treatment of Chronic Hepatitis B in Patients With Normal ALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Gilead Sciences (Industry); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-5944-A03
Record Dates: First submitted 2005-09-12; First posted 2005-09-30 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — adefovir dipivoxil; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mono therapy (Active Comparator): Hepsera
  Interventions: Drug: Hepsera
- Combo therapy (Active Comparator)
  Interventions: Drug: Hepsera and lamivudine

INTERVENTIONS:
Drug: Hepsera
  Arms: Mono therapy
Drug: Hepsera and lamivudine
  Arms: Combo therapy

SUMMARY:
This project is a randomized, open-label trial of adefovir dipivoxil (Hepsera) and lamivudine combination therapy versus adefovir dipivoxil (Hepsera) monotherapy. Both adefovir dipivoxil and lamivudine are nucleoside analogues approved by the U.S. FDA for the treatment of chronic hepatitis B.

The primary hypothesis is that subjects treated with combination therapy will see their viral DNA count decrease in an amount greater than subjects treated with monotherapy. The secondary hypothesis is that subjects treated with combination therapy will have a higher HBeAg conversion rate compared to historical controls of subjects treated with lamivudine or adefovir dipivoxil monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* HBsAg+ at screening and for at least 6 months prior to study entry
* HBeAg+
* HBV DNA greater than 6 log10 copies/mL
* Platelet count greater than 50,000 platelets/mm3
* Hemoglobin greater than 7.5 g/dL
* ALT less than ULN
* Estimated creatine clearance>50 mL/min as estimated by the Crockcroft-Gault equation ((140-age) x (kg)/(serum creatine x 72) (for women x 0.85))
* Female and male participants must be practicing an effective form of contraception (male or female condom with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, hormonal contraception)
* Serum alpha-fetoprotein less than 50 ng/mL within 30 days of study entry
* Childs-Pugh score less than 7 and no ascites, variceal bleeding, or hepatic encephalopathy
* able to give written informed consent and to comply with the study protocol

Exclusion Criteria:

* history or evidence of HIV, hepatitis C or hepatitis D
* known or suspected hypersensitivity to adefovir or other nucleoside/nucleotide analogs.
* history of clinically significant renal dysfunction
* any active medical or psychiatric illness that, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance with the protocol
* pregnancy or breastfeeding
* receipt of systemic corticosteroids within 90 days of study entry
* receipt of nephrotoxic drugs within 8 weeks prior to study screening or expected use of these agents during the course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Subjects treated with combination therapy will have a decrease in the viral DNA that is greater than the subjects treated with monotherapy. | one year

SECONDARY OUTCOMES:
Subjects treated with combination therapy will have an improved HBeAg conversion rate compared to historical controls treated with either lamivudine or adefovir dipivoxil monotherapy. | one year

CONTACTS AND LOCATIONS:
Overall Officials: John D Scott, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States